CLINICAL TRIAL: NCT01956084
Title: ADMINISTRATION of LMP-SPECIFIC CYTOTOXIC T-LYMPHOCYTES to PATIENTS with RELAPSED EBV-POSITIVE LYMPHOMA
Brief Title: Cytotoxic T Cells to Treat Relapsed EBV-positive Lymphoma
Acronym: ALCI2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Catherine Bollard (Other)
Responsible Party: Sponsor-Investigator, Catherine Bollard, Director- Program for Cell Enhancement and Technologies for Immunotherapy (CETI), Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALCI2
Record Dates: First submitted 2013-09-25; First posted 2013-10-08 (Estimated); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Hodgkin Disease; Non Hodgkin Lymphoma; Lymphoepithelioma; Severe Chronic Active EBV Infection Syndrome (SCAEBV); Leiomyosarcoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Leiomyosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- LMP1/2 CTLs (Group A) (Experimental): Patients receiving CTLs as adjunctive therapy following allogeneic stem transplant
  Interventions: Drug: LMP1/2 CTLs (Group A)
- LMP1/2 CTLs (Group B) (Experimental): Patients receiving CTLs in relapse following allogeneic stem cell transplant
  Interventions: Drug: LMP1/2 CTLs (Group B)

INTERVENTIONS:
Drug: LMP1/2 CTLs (Group A) — Each patient will receive 2 injections, 14 days apart, according to the following dosing schedules:
  Dose Level One:
  Day 0: 1 x 107 cells/m2 Day 14: 1 x 107 cells/m2
  Dose Level Two:
  Day 0: 2 x 107 cells/m2 Day 14: 2 x 107 cells/m2
  Dose Level Three:
  Day 0: 5 x 107 cells/m2 Day 14: 5 x 107 cells/m2
  Arms: LMP1/2 CTLs (Group A)
Drug: LMP1/2 CTLs (Group B) — Each patient will receive 2 injections, 14 days apart, according to the following dosing schedules:
  Dose Level One:
  Day 0: 1 x 107 cells/m2 Day 14: 1 x 107 cells/m2
  Dose Level Two:
  Day 0: 2 x 107 cells/m2 Day 14: 2 x 107 cells/m2
  Dose Level Three:
  Day 0: 5 x 107 cells/m2 Day 14: 5 x 107 cells/m2
  Arms: LMP1/2 CTLs (Group B)

SUMMARY:
In this study, investigators are trying to see if LMP specific cytotoxic T lymphocytes (CTLs) will prevent or treat disease called Epstein Barr Virus (EBV) Disorder including either Hodgkin Lymphoma or non-Hodgkin Lymphoma or Lymphoepithelioma or severe chronic active EBV infection syndrome (SCAEBV) or Leiomyosarcoma which has come back or has not gone away after treatment, including the best treatment. Investigators are using special immune system cells called third party LMP specific cytotoxic T lymphocytes (CTLs), a new experimental therapy.

Some patients with Lymphoma or SCAEBV or Leiomyosarcoma show evidence of infection with the virus that causes infectious mononucleosis Epstein Barr virus (EBV) before or at the time of their diagnosis. EBV is found in the cancer cells of up to half the patients with Hodgkin's and non-Hodgkin Lymphoma, suggesting that it may play a role in causing Lymphoma. The cancer cells (in lymphoma) and some B cells (in SCAEBV) infected by EBV are able to hide from the body's immune system and escape destruction. The investigators want to see if special white blood cells, called T cells, that have been trained to kill EBV infected cells can survive in patient's blood and affect the tumor or infection.

Investigators used this sort of therapy to treat a different type of cancer that occurs after bone marrow or solid organ transplant called post transplant lymphoma. In this type of cancer the tumor cells have 9 proteins made by EBV on their surface. They grew T cells in the laboratory that recognized all 9 proteins and were able to successfully prevent and treat post transplant lymphoma. However in Hodgkin Lymphoma, the tumor cells and B cells only express 2 EBV proteins. In a previous study they made T cells that recognized all 9 proteins and gave them to patients with Hodgkin Lymphoma. Some patients had a partial response to this therapy but no patients had a complete response. They think one reason may be that many of the T cells reacted with proteins that were not on the tumor cells. In this present study the investigators are trying to find out if the investigators can improve this treatment by growing T cells that recognize proteins expressed on EBV infected Lymphoma cells and B cells called LMP-1 and LMP2. These special T cells are called third party LMP 1/2 -specific cytotoxic T-lymphocytes (CTLs). These LMP-specific cytotoxic

T cells are an investigational product not approved by the Food and Drug Administration.

DETAILED DESCRIPTION:
Investigators will first test a biopsy of the tumor or lymph node that has already been done to see if the tumor or tissue cells are EBV positive. If the patient is eligible, investigators will then take 60 mL (about 12 teaspoons) of blood from the patient or their donor on one or two occasions. They will use this blood to grow T cells. First they will grow a special type of cells called dendritic cells or monocytes which will stimulate the T cells. Next they will put a specially produced human virus that carries the LMP genes into the dendritic cells or monocytes. They will then be used to stimulate T cells. This stimulation will train the T cells to kill cells with LMP on their surface. Investigators will then grow these LMP specific CTLs by more stimulation with EBV infected cells. These EBV infected cells will be treated with radiation so they cannot grow.

Once sufficient numbers of T cells have been made, investigators will test them to make sure they kill cells with LMP on their surface. If the counts are low they may need to obtain additional blood samples to make these cells. Prior to giving the patient the CTLs, the cells will be tested to make sure they don't attack the tissue.

The cells will then be thawed and injected into the patient over 10 minutes. Initially, two doses of T cells will be given two weeks apart. If after the second infusion there is a reduction in the size of the lymphoma on CT or MRI scan as assessed by a radiologist, the patient can receive up to six additional doses of the T cells if the patient wishes. This is a dose escalation study which means that for some patients the second dose may be larger than the first. All of the treatments will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital or the Methodist Hospital.

For follow-up after the CTL infusions, the patient will be seen every 3 months for the first year. Then the patient will either be seen in the clinic or they will be contacted by a research nurse yearly for 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient, regardless of age or sex, with a diagnosis of EBV positive Hodgkin's or non-Hodgkin's Lymphoma or EBV (associated)-T/NK-LPD lymphoproliferative disease or Lymphoepithelioma/leiomyosarcoma regardless of histological subtype or Severe Chronic EBV and in remission (group A) or with detectable disease (group B) after allogeneic SCT
2. Patients with life expectancy > 6 weeks.
3. Tumor tissue EBV positive
4. Patients with a Karnofsky/Lansky score of > 50
5. Donor HIV negative
6. must not have less than 50% donor chimerism in either peripheral blood or bone marrow
7. Patients with bilirubin <2x normal, AST <5x normal, and Hgb >8.0
8. Patients with a creatinine <2x normal for age
9. Patients should have been off other investigational therapy for one month prior to entry in this study.
10. Patient, parent/guardian able to give informed consent.

Exclusion Criteria:

1. Donors who are HIV positive
2. Patients with GVHD > Grade II
3. Due to unknown effects of this therapy on a fetus, pregnant women are excluded from this research.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-11; Primary Completion 2017-11-19 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicity (DLT) | 6 weeks
  Toxicity will be evaluated according to NCI Common Terminology Criteria for Adverse Events scale, version 2.0. DLT will be defined as development of any toxicity scored as Grade 3 or 4 and primarily related to the CTL infusion.

SECONDARY OUTCOMES:
Survival and Immune Function of LMP-specific CTLs | 5 years
  Survival and function will be measured by frequencies and immunological parameters from (enzyme-linked immunospot) ELISPOT and cytotoxicity assays.

OTHER OUTCOMES:
To obtain preliminary information on the safety and response to an extended dosage regimen. | 6 weeks
  Comparison of diagnostic imaging studies from pre-infusion to 6 weeks after the second infusion will be summarized. Frequencies and proportions of responders will be summarized overall and by dose levels if there are enough patients per dose level.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Bollard, MD, Principal Investigator — CNMC
Locations (1):
- Childrens National Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] McLaughlin LP, Rouce R, Gottschalk S, Torrano V, Carrum G, Wu MF, Hoq F, Grilley B, Marcogliese AM, Hanley PJ, Gee AP, Brenner MK, Rooney CM, Heslop HE, Bollard CM. EBV/LMP-specific T cells maintain remissions of T- and B-cell EBV lymphomas after allogeneic bone marrow transplantation. Blood. 2018 Nov 29;132(22):2351-2361. doi: 10.1182/blood-2018-07-863654. Epub 2018 Sep 27. PMID 30262660